CLINICAL TRIAL: NCT05592392
Title: RECOVER-HF Pilot Study - Randomized, Single-Center, Double-blinded Study of Synchronized Diaphragmatic Stimulation (SDS) for Improvement of Symptomatic Reduced Ejection Fraction Heart Failure
Brief Title: RECOVER-HF Pilot Study of SDS in Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VisCardia Inc. (Industry)
Collaborators: Clinical Accelerator (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: VisCardia H02_22
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Heart Failure; Heart Disease; Cardiovascular Diseases; Synchronized Diaphragmatic Stimulation; Implantable Heart Failure Device Therapy
MeSH Terms: conditions — Heart Failure; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Partial crossover - initial randomized to therapy On/Off. Subsequent OFF converted to On after primary efficacy endpoint.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Investigator blinded to device programming, therapy imperceptible to patient
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapy (Experimental): SDS system implanted and Therapy On for 6 months post randomization
  Interventions: Device: Synchronized Diaphragmatic Stimulation
- Control (Sham Comparator): SDS system implanted and Therapy Off for 6 months post randomization
  Interventions: Device: Synchronized Diaphragmatic Stimulation

INTERVENTIONS:
Device: Synchronized Diaphragmatic Stimulation — Implantable Pulse Generator system providing cardiac-gaited stimulation of the diaphragm and thereby influence cardiovascular properties relevant in heart failure.
  Other Names: ADS, SDS, VisONE SDS

SUMMARY:
The RECOVER HF pilot is a feasibility study for evaluating a randomized, doubled-blinded study design to determine the benefits and risks of chronically delivering Synchronized Diaphragmatic Stimulation (SDS) in Heart Failure patients on GDMT with NYHA II/III, EF<=40% and QRSd,=130ms.

DETAILED DESCRIPTION:
Symptomatic Diaphragmatic Stimulation (SDS) is a novel approach designed to improve cardiac function, symptoms, and, ultimately, outcomes for patients who are symptomatic for heart failure.

Elevated intracardiac pressures are the hallmark of heart failure (HF) and a key pathological driver of disease progression and limited exertional capacity. The degree of cardiac pressure elevation is determined by preload, afterload, and pericardial restraint. The pericardium restrains the heart, and the degree of restraint is determined by the pericardial structure itself and the intrathoracic pressure. This aspect of HF pathophysiology is among the fundamental drivers behind the SDS therapy concept. SDS induces a temporal modulation of intrathoracic pressure with a resultant reduction in pericardial restraint, leading to improved cardiac filling and reduced afterload. When applied at the right time in the cardiac cycle, SDS can improve cardiac filling, cardiovascular pressure conditions, and systolic cardiac performance.

Encouraged by the results of the VisONE HF study pilot (NCT03484780), SDS shall now be further valuated in a randomized controlled trial (RCT) pilot. This RCT pilot has three objectives: two semi-acute items (15-30 days) verification of sensing function using the modified input filters and improved usability based on increased automaticity of the user-interface; and one chronic result (6 months) to reproduce similar efficacy endpoints. The herein described study is a pilot trial for a larger RCT trial.

ELIGIBILITY:
Inclusion Criteria:

* NYHA classes II/III on optimal Guideline Directed Medical Therapy
* QRS duration ≤ 130 ms
* LVEF < 40%
* Willing and able to comply with protocol requirements, including attending all required visits
* Wiling to participate in the study and able to sign an informed consent form

Exclusion Criteria:

* Baseline 6-minute walk test > 500 meters or < 200 meters
* NT-proBNP< 250 if on loop diuretics, or NT-proBNP < 500 if not on loop diuretics
* Supine resting heart rate > 140 bpm
* Systolic blood pressure < 80 mmHg or > 170 mmHg
* Serum creatinine > 2.5 mg/dL
* Serum hepatic function 3x ULN
* Unstable angina, AMI, CABG, PTCA, CVA/TIA, persistent AF, NSVT or DCCV within 3 months
* Intermittent IV inotropic drug treatment
* Arrhythmias present during screening (profound ectopy, bradycardia, profound prevalence of ectopy, NSVT, VF, AF*, SVT or AFLT) - * see enrollment exception allowing for 10 patients in AF for a separate subgroup analysis
* Reversible non-ischemic cardiomyopathy
* Primary valvular disease
* Severe primary pulmonary disease, including pulmonary arterial hypertension. PAP sys >70 mmHg at rest
* Severe COPD, other respiratory or lung diseases where FEV < 50%
* Pericardial disease
* Diabetic neuropathy
* Existing diaphragmatic stimulation for respiration assist
* LVAD or other mechanical cardiac assist devices
* Contraindications to laparoscopic access to the diaphragm, as determined by the implanting physician
* Known intra-abdominal pathology which could increase the risk of laparoscopic access to the diaphragm.
* Previous open laparotomy within 1 year
* Previous thoracic or abdominal organ transplant
* Drug induced immuno-suppression
* Body mass index > 40
* Enrollment in a concurrent investigation / clinical study
* Having a life expectancy of <1 year due to any condition
* Pregnant or planning a pregnancy during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Change in LVESV | 6 months
  Change from baseline in left ventricular end systolic volume (LVESV) post-randomization between the control group and the therapy group.
Freedom from VisONE device-related and procedure-related Major Adverse Respiratory and Cardiovascular Events (MARCE) after the index implantation procedure | 12 months
  The following Major Respiratory and Cardiovascular Events will be analyzed for their rate and severity and association with the implantable device or procedure:
  1. CV Death
  2. Stroke
  3. Cardiac Arrest
  4. Interaction with cardiac rhythm device requiring permanent termination of SDS therapy
  5. Acute Heart Failure Decompensation
  6. Infection requiring device/lead explant
  7. Diaphragmatic dysfunction leading to a clinically significant reduction is respiratory function
  8. Inadequate SDS therapy delivery requiring surgical intervention
  9. Injury to abdominal organs requiring surgical intervention
  10. Pneumothorax
  11. Hemothorax
  12. Peritonitis

SECONDARY OUTCOMES:
Change in 6MHW distance | 6 months
  Change from baseline in 6 MHW distance post-randomization between the control group and the therapy group.
Change in MLWHF overall score | 6 months
  Change from baseline in MLWHF total score post-randomization between the control group and the therapy group.

CONTACTS AND LOCATIONS:
Overall Officials: Tamaz Shaburishvili, MD, PhD, Principal Investigator — Tbilisi Heart and Vascular Clinic
Locations (2):
- Tbilisi Heart And Vascular Clinic, Tbilisi, Georgia
- Republican Specialized Scientific and Practical Medical Center for Surgery n.a. V. Vakhidov, Tashkent, Uzbekistan

IPD SHARING:
Plan to Share IPD: No